CLINICAL TRIAL: NCT01048398
Title: Remifentanil Versus Placebo for Pain Treatment External Cephalic Versions. Randomized, Controlled and Masked
Brief Title: Remifentanil Versus Paracetamol for Pain Treatment External Cephalic Versions.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Cesar Augusto Valero Martinez, Hospital Txagorritxu
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REMI-001
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2010-09

CONDITIONS: Breech Presentation; Pregnancy
Keywords: ceophalic version; breech presentation; pregnancy; remifentanil; paracetamol
MeSH Terms: conditions — Breech Presentation | interventions — Remifentanil; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentanil (Experimental)
  Interventions: Drug: remifentanil
- Paracetamol (Active Comparator): intravenous paracetamol 1g
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: remifentanil — intervention: intravenous paracetamol 1g and remifentanil 1mg/100ml in 100ml of 0.9% saline.
  Arms: Remifentanil
Drug: paracetamol — Control group: intravenous paracetamol 1g
  Other Names: acetoaminophen
  Arms: Paracetamol

SUMMARY:
BACKGROUND: Between 3-4% of pregnancies carried to term, the fetuses are in breech presentation. The external version is a maneuver gynecological used to turn a breech in cephalic presentation. For treatment of pain suggests the use of μ agonist remifentanil for fast action and elimination.

OBJECTIVE: To compare the effectiveness of remifentanil for pain management in external version.

PATIENTS: Pregnant for 36 weeks or more with breech presentation who met the inclusion criteria and sign the consent. Participants will be randomized into two groups before the procedure.

Group intervention: paracetamol and remifentanil Control group: paracetamol and placebo DETERMINATIONS: VAS pain level, percentage of success of the maneuver and adverse events.

Statistical Analysis: Comparison of pain recorded by VAS in both groups and comparison of adverse events

ELIGIBILITY:
Inclusion Criteria:

* Fetuses between weeks 36 and 41 of gestation confirmed by ultrasound with non-cephalic presentation.
* Informed consent signed by the mother or legal representative in his absence.

Exclusion Criteria:

* Fetal anomalies
* Severe hypertension
* Allergy to drug used in the test
* Amniotic fluid index ≥ 5 cm
* Contraindication for vaginal delivery
* Uterine abnormality and impaired coagulation
* Placenta previa
* Rh sensitization
* Multiple gestation
* Ruptured membranes
* Premature detachment of normally inserted placenta
* The mother greater weight to 85kg

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Degree of decrease in pain experienced by patients during the maneuver according to the VAS | 10 minutes

SECONDARY OUTCOMES:
Proportion of patients in each group in which the procedure is effective and avoids performing a Caesarean section. | 1 day
Number of adverse events and severity | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Cesar A Valero, MD, Principal Investigator — Basque Health Service; Henar Muñoz, MD, Study Chair — Basque Health Service; Amanda Lopez, Study Chair — Basque Health Service; Sandra Guerra, MD, Study Chair — Basque Health Service; Olga Echebarria, MD, Study Chair — Basque Health Service; Alfonso Velasco, MD, Study Chair — University of Valladolid
Locations (1):
- Hospital Txagorritxu, Vitoria-Gasteiz, Alava, Spain